CLINICAL TRIAL: NCT05119868
Title: Effects of the Mediterranean Diet During Pregnancy on the Onset of Allergies in the Offspring: a Multi-center Randomised-controlled Trial (the PREMEDI Project)
Brief Title: Effects of the Mediterranean Diet During Pregnancy on the Onset of Allergies in the Offspring
Acronym: PREMEDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Professor of Pediatrics, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 283/21
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-06

CONDITIONS: Allergies; Obesity; Gestational Complications; Gestational Weight Gain; Perinatal Condition; Birth Weight; Chronic Diseases in Children; Breast Feeding
MeSH Terms: conditions — Hypersensitivity; Obesity; Gestational Weight Gain; Birth Weight; Breast Feeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will receive standard obstetrical and gynecological follow-up and nutritional intervention based on Mediterranean Diet provided by certified dietitians
  Interventions: Other: Nutritional intervention based on Mediterranean Diet
- Group 2 (No Intervention): Group 2 will receive standard obstetrical and gynecological follow-up alone

INTERVENTIONS:
Other: Nutritional intervention based on Mediterranean Diet — A personalized nutritional counseling and a tailored diet, according to Mediterranean dietary pattern, designed on the pre-pregnancy weight, height and trimester of pregnancy provided by certified dietitians.
  Arms: Group 1

SUMMARY:
Allergy prevalence is increasing steadily with some describing as the "epidemic of the twenty-first century". Maternal diet during pregnancy has been linked to offspring allergy risk, so it represents a potential target for allergy prevention. The Mediterranean Diet (MD) is considered one of the healthiest dietary models which exerts regulatory effects on immune system, due to the synergistic and interactive combinations of nutrients. We aim to study the effects of MD in pregnancy on the onset of allergic diseases at 2 years of age in the offspring.

ELIGIBILITY:
Inclusion Criteria:

- healthy women (aged 20-35 years), at first trimester of pregnancy, of at risk for atopy baby

Exclusion Criteria:

* concomitant presence of infections;
* concomitant presence of malignancies;
* concomitant presence of major gastrointestinal malformations;
* concomitant presence of immunodeficiencies;
* concomitant presence of autoimmune diseases;
* concomitant presence of chronic inflammatory bowel diseases;
* concomitant presence of functional gastrointestinal disorders;
* concomitant presence of celiac disease;
* history of abdominal surgery with gastrointestinal resection;
* concomitant presence of neuropsychiatric disorders;
* concomitant presence of central nervous system disorders;
* vegan diet;
* twin pregnancy;
* concomitant presence of genetic disorders;
* concomitant presence of metabolic disorders.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of allergic disorders at 24 months of age in the offspring | 24 months from birth
  The evaluation of the effect of Mediterranean Diet during pregnancy on the occurrence of allergic disorders at 24 months of age in the offspring

SECONDARY OUTCOMES:
Maternal weight gain | From enrollment until delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on maternal weight gain
Pregnancy complications occurrence | From enrollment until delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on pregnancy complications occurrence
Perinatal complications occurrence | Delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on perinatal complications occurrence
Neonatal birth weight | Delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on neonatal growth indices
Body growth in the offspring | During the 24 months of life
  The evaluation of the effect of Mediterranean Diet during pregnancy on body growth in the offspring
Occurrence of any other chronic disorders in the first 2 years of age in the offspring | During the 24 months of life
  The evaluation of the effect of Mediterranean Diet during pregnancy on the occurrence of any other chronic disorders in the first 2 years of age in the offspring
Mother's gut microbiome metagenomic features | From enrollment until delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on the mother's gut microbiome metagenomic features
Mother's gut microbiome metabolomic features | From enrollment until delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on the mother's gut microbiome metabolomic features
Son's gut microbiome metagenomic features | During the 24 months of life
  The evaluation of the effect of Mediterranean Diet during pregnancy on the son's gut microbiome metagenomic features
Son's gut microbiome metabolomic features | During the 24 months of life
  The evaluation of the effect of Mediterranean Diet during pregnancy on the son's gut microbiome metabolomic features
Breastfeeding duration | During the 24 months of life
  The evaluation of the effect of Mediterranean Diet during pregnancy on the breastfeeding duration
Breast milk composition | During the 24 months of life
  The evaluation of the effect of Mediterranean Diet during pregnancy on the breast milk composition
Epigenetic modulation of genes involved in the regulation of immune system in the offspring | Delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on the epigenetic modulation of genes involved in the regulation of immune system in the offspring
Epigenetic modulation of genes involved in the metabolic pathways in the offspring | Delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on the epigenetic modulation of genes involved in the metabolic pathways in the offspring
To validate a digital app | During the first 1000 days
  Validate an app designed to promote a healthy lifestyle and prevent the most common non-communicable chronic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, Principal Investigator — Department of Traslational Medical Science at University of Naples Federico II
Locations (2):
- Italy (2):
  - Department of Traslational Medical Science - University of Naples Federico II, Naples
  - Department of Traslational Medical Science, Naples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coppola S, Paparo L, Chiariotti L, Ercolini D, Nocerino R, de Giovanni di Santa Severina AF, Carucci L, De Filippis F, Agangi A, Napolitano M, Passariello A, Messina F, Berni Canani R. Effects of the Mediterranean Diet during pregnancy on the onset of allergy in at risk children: A study protocol of a multi-center, randomized- controlled, parallel groups, prospective trial (the PREMEDI study). Front Nutr. 2022 Oct 13;9:951223. doi: 10.3389/fnut.2022.951223. eCollection 2022. PMID 36313083